CLINICAL TRIAL: NCT06096415
Title: A Parallel Group Treatment, Phase 2A, Double-blind, 3-arm Study to Investigate Safety and Efficacy of ABX-101 Compared With Placebo in Male and Female Participants, Aged 18 to 50 Years, With Moderate-to-severe Traumatic Brain Injury
Brief Title: Safety and Efficacy of ABX-101 in Participants Aged 18 to 50 Years of Age With Moderate to Severe Traumatic Brain Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abalonex, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABX-TBI-001
Record Dates: First submitted 2023-05-02; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Traumatic Brain Injury; Cerebral Edema
Keywords: Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Edema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: ABX-101 1mg (Experimental): Participants will be screened, enrolled and receive the assigned treatment within 12 hours of the primary TBI insult (or estimated less than 12 hours if the exact time is unknown).
  Enrolled participants will be stratified 1:1 (in each arm) by GCS score (GCS 4-8 in one group and GCS 9 - 12 in the other).
  The treatment period, which involves 6 hourly, i.e., quarter in die (QID), ABX 101 (1 mg OR 2 mg) intramuscular injections, is seven days.
  Interventions: Drug: ABX-101 1mg; Drug: ABX-101 2mg
- Experimental: ABX-101 2mg (Experimental): Participants will be screened, enrolled and receive the assigned treatment within 12 hours of the primary TBI insult (or estimated less than 12 hours if the exact time is unknown).
  Enrolled participants will be stratified 1:1 (in each arm) by GCS score (GCS 4-8 in one group and GCS 9 - 12 in the other).
  The treatment period, which involves 6 hourly, i.e., quarter in die (QID), ABX 101 (1 mg OR 2 mg) intramuscular injections, is seven days.
  Interventions: Drug: ABX-101 1mg; Drug: ABX-101 2mg
- Placebo Comparator: Saline (Placebo Comparator): Placebo to the ABX-101 will be administered to patients.
  Interventions: Drug: ABX-101 1mg; Drug: ABX-101 2mg

INTERVENTIONS:
Drug: ABX-101 1mg — ABX-101 1mg will be provided to patients stratified 1:1 by GCS scoring (GCS 4-8; GCS 9-12)
Drug: ABX-101 2mg — ABX-101 2mg will be provided to patients stratified 1:1 by GCS scoring (GCS 4-8; GCS 9-12)

SUMMARY:
The purpose of this study is to investigate the clinical improvement measured by the Glasgow Outcome Scale Extended (GOS-E) with ABX-101 compared with Placebo intramuscular injection in participants with moderate to severe TBI.

DETAILED DESCRIPTION:
Study details include:

* The study duration will be up to 180 days per participant.
* The treatment duration will be up to 7 days.
* The visits post-treatment will be on day 30 and day 180 of the study.

Number of Participants:

A maximum of 45 participants will be enrolled into the study and randomized to each treatment arm in a ratio of 1:1:1. i.e., fifteen participants per arm.

Study Arms and Duration:

Participants will be screened, enrolled and receive the assigned treatment within 12 hours of the primary TBI insult. Enrolled participants will be stratified 1:1 (in each arm) by GCS score (GCS 4-8 in one group and GCS 9 - 12 in the other). The treatment period, which involves 6 hourly, i.e., quarter in die (QID), ABX-101 (1 mg OR 2 mg) intramuscular injections, is seven days. Enrolled participant will continue with the in-hospital standard of care, as decided by the external treating physician, and will be followed up by the study team on days 30 and days 180. The ABX-101 1 mg and 2 mg arm will be enrolled simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from patient, patient's legal guardian or legal representative, or deferred consent procedure, according to local requirements
* 18 - 50 years of age, inclusive
* Expected to survive more than 24 hours after admission
* Clearly defined time of injury no more than 12 hours before administration of study drug/placebo

  o Subjects stratified 1:1 (in each arm) by treatment administered 0-12 hrs
* TBI with Glasgow Coma Score (GCS) 4-12 requiring intracranial pressure (ICP) monitoring according to the assessment of the treating physician

  o Subjects stratified 1:1 (in each arm) by GCS 4-8 and GCS 9-12
* Catheter placement (intraventricular or intraparenchymal, only) for monitoring and management of increased ICP
* [Brain computed tomography (CT) showing intracranial parenchymal abnormality and hemodynamically stable]

Exclusion Criteria:

* Penetrating head injury (e.g. missile, stab wound)
* Concurrent, but not pre-existing, spinal cord injury
* Not expected to survive more than 24 hours after admission
* Pregnant, or a positive pregnancy test
* Coma due to an exclusive epidural hematoma (lucid interval and absence of structural brain damage on CT scan)
* Patient pupils are unresponsive (dilation) in both eyes
* The subject has a neurodegenerative disease or other neurological disorder including dementia, Parkinson's disease, multiple sclerosis, seizure disorder, or brain tumors.
* Coma suspected to be primarily due to other causes than head injury (e.g. drug overdose intoxication, drowning/near drowning
* Known or CT scan evidence of pre-existing major cerebral damage
* Any severe concomitant condition (cancer; hematologic, renal, hepatic, coronary disease; major psychiatric disorder; alcohol or drug abuse), that can be ascertained at admission
* Known to have received an experimental drug within 4 weeks prior to current injury
* Patients who cannot be monitored with regard to their recovery (GOS-E and QOLIBRI)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale-Extended (GOS-E) | 180 days
  To demonstrate superiority of ABX-101 vs placebo on the Glasgow Outcome Scale-Extended (GOS-E) at 90-days in participants with TBI

SECONDARY OUTCOMES:
Glasgow Outcome Scale-Extended (GOS-E) | 30 days
  To demonstrate superiority of ABX-101 vs placebo on the GOS-E at 30 days in participants with TBI
Glasgow Coma Score (GSC) improvement | 7 days
  To demonstrate superiority of ABX-101 vs placebo on the GCS improvement (vs. baseline) at days 3 and 7 in participants with TBI
ICP Maintenance | 7 days
  To demonstrate superiority of ABX-101 vs placebo on the ICP maintenance at 3 days and 7 days in participants with TBI
Midline Shift | 3 days
  To demonstrate superiority of ABX-101 vs placebo on the degree of midline shift as assessed by CT scan at 1 day and 3 days in participants with TBI
Therapeutic Intensity Level | 7 days
  To demonstrate superiority of ABX-101 vs placebo on the Therapeutic Intensity Level over 3 days and over 7 days in participants with TBI
Neuroworsening | 7 days
  To demonstrate superiority of ABX-101 vs placebo on the Neuroworsening at 3 days and 7 days in participants with TBI
Mortality | 180 days
  To demonstrate superiority of ABX-101 vs placebo on the mortality at 3 days, 7 days, 28 days, and 90 days in participants with TBI
Quality of life- (QOLIBRI) | 180 days
  To demonstrate superiority of ABX-101 vs placebo on the Quality of Life after Brain Injury at 90 days in participants with TBI
GFAP Inflammatory Biomarker Analysis | 7 days
  To compare ABX-101 vs placebo on Glial fibrillary acidic protein (GFAP) levels at 1 day, 3 days, and 7 days in participants with TBI. The detection range for GFAP biomarker is 0.31 - 20 ng/ml using ELAB Science GFAP Kit.
Adverse Events | 7 days
  To compare ABX-101 vs placebo in terms of AEs assessed over 7 days of treatment and through the duration of follow-up in participants with TBI